CLINICAL TRIAL: NCT06853002
Title: Comparison Between Deep Breathing Exercises and Incentive Spirometry After Rib Fracture
Brief Title: Deep Breathing Exercises and Incentive Spirometry After Rib Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GOKAEK 2025/2/2
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-02

CONDITIONS: Rib Fractures; Oxygenation
Keywords: Rib Fractures; Breathing exercises; Postoperative complications
MeSH Terms: conditions — Rib Fractures; Postoperative Complications | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Active Comparator): Spirometer group
  Interventions: Other: Breathing exercise with spirometry
- Group D (Active Comparator): Deep breathing exercise group
  Interventions: Other: Breathing exercise with deep breathing method

INTERVENTIONS:
Other: Breathing exercise with spirometry — Breathing exercise with spirometry
  Arms: Group S
Other: Breathing exercise with deep breathing method — Breathing exercise with deep breathing method
  Arms: Group D

SUMMARY:
Chest trauma patients constitute approximately 10-15% of all traffic accidents. Many complications may occur after chest trauma, including rib fracture, pneumothorax, hemothorax, lung contusion, flail chest, atelectasis, respiratory failure and even death. Atelectasis is the most common of these complications. This study planned to investigate the effects of spirometry and deep breathing exercises on oxygenation after rib fracture.

DETAILED DESCRIPTION:
Chest trauma is the second leading cause of death in traffic accidents, accounting for approximately 25% of deaths, only slightly lower than deaths from head injuries. Chest trauma can involve various organs, including the heart, great vessels, lungs, trachea, and esophagus or chest wall. Complications of rib fractures can follow, including pneumothorax, hemothorax, pulmonary contusion, flail chest, atelectasis, respiratory failure, and even death. Atelectasis is the most common complication. Patients with rib fractures usually do not require surgical intervention. However, hospitalization for pain control and further observation is necessary to maintain lung hygiene and prevent further complications. Patients with rib fractures usually complain of chest pain due to impaired lung hygiene, obstruction of the lower airway, and subsequent atelectasis and hypoventilation. Hypoxemia, pneumonia, respiratory failure, and other morbidities can lead to prolonged hospital stays and mortality.

spirometry exercise and deep breathing exercises are breathing exercises that help expand the lungs. They are often used to prevent postoperative lung atelectasis and reduce pulmonary complications after cardiac, lung, or abdominal surgery. They can increase maximum inspiratory capacity and lung compliance, improve oxygenation, and maintain lower airway patency to prevent and treat atelectasis.

Patients admitted to the intensive care unit due to rib fractures will be randomized into two groups according to the closed envelope drawing method. (Group S: spirometry group, Group D: deep breathing exercise group). Patients over the age of 18 who developed rib fractures due to thoracic trauma will be included in the study. Demographic characteristics, trauma score, systemic diseases, presence of lung contusion, number of rib fractures, additional trauma status laboratory values of the patients will be recorded.

The pain level of the patients will be monitored with Numeric rating scale (NRS) and the target will be NRS:0-2. The analgesia regimen will be recorded for this purpose.

Group S: Spirometry exercises will be performed in a sitting position by holding the device, exhaling normally and then closing the lips tightly around the mouthpiece. Then, the patient will perform maximum inspiration by taking long, deep and slow breaths. When the patient takes a deep breath, the balls in the chamber rise, after maximum inhalation, the patient will be asked to hold their breath for 3-5 seconds, then remove the mouthpiece and exhale slowly. spirometry exercises will be prescribed daily for follow-up in the intensive care unit, five times a day, ten repetitions each, with 1-2 hours of rest between exercises.

Group D: The patient will be asked to sit in a comfortable position with their hands on their lap, press the tip of their tongue to the tissue behind their upper front teeth and hold it there throughout the breathing cycle. After three normal breaths, they will take a deep breath through the nose for 4 counts, hold their breath for 7 counts, and then exhale slowly through the mouth for 8 counts and repeat the breathing cycle. This cycle will be applied five times a day, ten repetitions, during the follow-up in the intensive care unit.

The effect of these practices on oxygenation will be evaluated according to saturation and routine blood gas results.

In this study, the effects of spirometry and deep breathing exercises on oxygenation after rib fracture will be investigated as the primary objective, and the effects of spirometry and deep breathing exercises on the duration of intensive care stay will be investigated as the secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed rib fractures due to thoracic trauma

Exclusion Criteria:

* Patients who are unconscious
* Patients with a history of chronic obstructive pulmonary disease or asthma
* Patients with an Injury Severity Score (ISS) ≥ 16
* Patients who require mechanical ventilation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Breathing exercise in rib fractures | 3 day
  Comparison of the effects of spirometry and deep breathing exercise on oxygenation levels in patients with rib fractures

SECONDARY OUTCOMES:
Breathing exercise on intensive care unit time | 7 days
  Effect of respiratory exercise on intensive care unit time in patients with rib fractures

CONTACTS AND LOCATIONS:
Overall Officials: özgür kömürcü, Study Director — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renault JA, Costa-Val R, Rosseti MB, Houri Neto M. Comparison between deep breathing exercises and incentive spirometry after CABG surgery. Rev Bras Cir Cardiovasc. 2009 Apr-Jun;24(2):165-72. doi: 10.1590/s0102-76382009000200012. PMID 19768295
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Hu L, Hua Y, Wang L, Mao Z, Jia X, Lei Z, Chang D, Cheng W. Effect of Short-term Deep Breathing Exercises on Perioperative Anxiety and Pain in Pediatric Orthopedic Patients: A Randomized Controlled Trial. J Perianesth Nurs. 2025 Feb;40(1):69-75. doi: 10.1016/j.jopan.2024.03.009. Epub 2024 Jul 9. PMID 38980240